CLINICAL TRIAL: NCT05622500
Title: Best Endovenous Treatment, Including STenting, Versus Non-endovenous Treatment in Chronic Proximal Deep Venous Disease - the BEST Multi-centre Randomised Controlled Trial
Brief Title: Best Endovenous Treatment, Including STenting, Versus Non-endovenous Treatment in Chronic Proximal Deep Venous Disease
Acronym: BEST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial failed to meet the milestones in the internal pilot of feasibility. The trial was redesigned to improve its deliverability and reduce burden to sites prior to being relaunched. Unfortunately, the trial failed to sufficiently recruit.
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22SM7477
Record Dates: First submitted 2022-11-07; First posted 2022-11-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Chronic Venous Insufficiency; Chronic Venous Thrombosis; Iliac Vein Stenosis; Iliac Vein Obstruction; Post Thrombotic Syndrome
Keywords: Deep venous stenting; Intravascular ultrasound; Post thrombotic syndrome; Non-thrombotic iliac vein lesions; Proximal venous outflow obstruction; Chronic venous disease
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Intervention Model Description: Superiority comparison using intention to treat analysis
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor-blinded (single blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best endovenous reconstruction + best medical treatment (compression +/- anti-thrombotic therapy). (Experimental): The intervention arm consists of participants undergoing best endovenous reconstruction under the guidance of intra-vascular ultrasound in addition to best medical treatment (compression +/- antithrombotic therapy).
  Interventions: Procedure: Deep venous stenting; Combination Product: Best medical therapy
- Best medical treatment alone (compression +/- anticoagulation). (Active Comparator): The comparator arm will consist of participants receiving best medical treatment alone.
  Interventions: Combination Product: Best medical therapy

INTERVENTIONS:
Procedure: Deep venous stenting — Endovascular reconstruction encompasses balloon venoplasty and venous stenting. A dedicated venous stent will be used, the brand of which the individual interventionist will decide.
  Other Names: Deep venous reconstruction; Iliac vein stenting
  Arms: Best endovenous reconstruction + best medical treatment (compression +/- anti-thrombotic therapy).
Combination Product: Best medical therapy — Compression stockings encompass a range of therapies used to provide an externally applied graduated-pressure up the length of the limb aiming to improve venous function and decrease lower limb swelling. Compression stockings can be classified by size and grade, i.e. the pressure the stockings applies to the limb. For the purpose of this trial Class II and Class III graduated compression stockings should be used, with the aim of providing Class III if tolerated. Antithrombotic agents include, but are not limited to: warfarin (titrated to international normalised ratio, INR), apixaban, rivaroxaban, aspirin, and clopidogrel.

SUMMARY:
Chronic obstruction of the iliac veins or inferior vena cava can occur as a result of deep vein thrombosis (DVT), or due to extrinsic compression in non-thrombotic iliac vein lesions (NIVLs). This obstruction can manifest as post-thrombotic syndrome (PTS) after DVT or as chronic venous disease (CVD) in NIVL. Despite sparse evidence, rates of venous stenting for PTS and NIVLs are increasing.

A pragmatic, observer-blind, multi-centre, randomised-controlled trial for adults with CVD secondary to either PTS or NIVLs randomised to either best endovenous therapy (including venoplasty and deep venous stenting) or standard therapy (compression +/- anticoagulation). Included participants will have chronic venous disease (CEAP classification 3 - 6) secondary to proximal deep venous disease. The primary outcome is severity of venous disease at 6 months as ascertained by the Venous Clinical Severity Score (VCSS).

DETAILED DESCRIPTION:
Symptomatic chronic obstructive lesions of the iliac veins and inferior vein cava can be secondary to post-thrombotic lesions caused by a deep vein thrombosis (DVT) or due to non-thrombotic iliac vein lesions (NIVLs). DVT has an annual incidence of 148 per 100,000 person years in Europe. Following a DVT, up to 50% of patients develop post thrombotic syndrome (PTS), defined as "chronic venous symptoms or signs secondary to DVT" i.e. lifelong leg pain, oedema and skin changes. Furthermore, the subsequent rate of venous ulceration is high with up to 29% of those with PTS suffering from active or healed venous ulcers. The pathophysiology of PTS is thought to be sustained venous hypertension from a combination of venous outflow obstruction and valvular incompetence. NIVLs are due to external compression or intrinsic lesions that reduce the venous drainage through the iliac venous system. This, in turn, can lead to chronic venous insufficiency and also increase the risk of DVT. NIVLs contribute to the significant morbidity and cost associated with CVD. NIVLs can be demonstrated on imaging as a stenosed iliac vein or in an iliac vein of normal diameter with intrinsic lesions.

Rates of venous stenting for PTS and NIVLs are rapidly increasing. However, sparse evidence exists to support the use of venous stenting and clinical guidelines reflect this. Endovenous stenting is being increasingly used as a treatment option for individuals with complications relating to chronic venous disease such as skin changes, ulceration, debilitating symptoms, and functional impairment. However, a recent systematic review of sixteen eligible studies, none of which were RCTs, concluded that: "The quality of evidence to support the use of deep venous stenting to treat chronic obstructive disease is currently weak. The treatment does however appear promising and is safe and should therefore be considered as a treatment option while the evidence base is improved". Many of the studies employed stents which were not primarily designed for use in the venous system. The role of endovenous reconstruction in the context of patients with PTS and NIVLs, including deep venous stenting using modern stents designed specifically for use in the venous system, remains to be elucidated in a well-designed RCT.

The rational for the proposed study is supported by both haemodynamic and clinical evidence. Retrospective cohorts of deep venous stenting in PTS and NIVLs have yielded promising results. Pre-clinical research suggests that common femoral vein pressure is increased in post thrombotic venous obstruction. It has been demonstrated that deep venous stenting improves mean ambulatory venous pressures and therefore should reduce the symptomology experienced by the individual. Furthermore, venous stents are specifically designed to be uncovered and rigid, aiming to keep the aspect ratio of the stent at a 1:1 ratio, to minimise outflow obstruction and increase venous return.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with chronic venous disease secondary to chronic proximal thrombotic or nonthrombotic stenosis or occlusion
2. Disease in iliac and/or caval deep venous system(s)
3. CEAP clinical C3, C4, C5, C6 or symptoms of venous claudication
4. Anatomically suitable for endovenous reconstruction

Exclusion Criteria:

1. Contraindications to stenting (e.g. anatomically unsuitable, contrast allergy)
2. Contraindications to prolonged anticoagulation
3. Existing diagnosis of profound pro-thrombotic states (Beh et's, anti-phospholipid syndrome)
4. Caval occlusion at or proximal to the level of the renal veins
5. Open / hybrid open-endovascular deep venous intervention
6. Pregnancy
7. Inability to provide consent
8. Need to intervene caudal to common femoral vein confluence to achieve inflow
9. Participants that have tested positive for coronavirus within the last 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Venous Clinical Severity Score (VCSS) at 6 months | 6 months
  Disease severity score. Venous clinical severity score (VCSS) encompasses nine hallmarks of chronic venous disease, each scored on a severity scale from 0 to 3. Min score 0, Max score 30. High score = worse severity of disease.

SECONDARY OUTCOMES:
Re-intervention, number of participants requiring an additional procedure. | 6 weeks, 3 months, 6 months, 12 months
  Dichotomous outcome, defined as additional procedure undertaken to maintain or re-establish stent patency,
Stent patency, dichotomous outcome, number of participants with a patent stent at last follow-up. | 6 weeks, 3 months, 6 months, 12 months
  Reported as primary, primary-assisted, secondary patency
Cost-effectiveness of deep venous reconstruction | 12 months
  ICER
VEINES-QoL/Sym | 6 weeks, 6 months, 12 months
  Disease-specific quality of life measure. Standardised score, hence no meaningful min/max. High score = better quality of life.
Villalta score | 6 weeks, 6 months, 12 months
  Disease severity score. Min score 0, Max score 33. High score = worse severity of disease.
Ginsberg score, dichotomous outcome (Yes / No) | 6 weeks, 6 months, 12 months
  Diagnostic system for PTS (Yes /No).
Venous ulceration, dichotomous outcome | 6 weeks, 6 months, 12 months
  Presence of venous ulceration on clinical examination.
SF-36 | 6 weeks, 6 months, 12 months
  Quality of life measure. Standardised score, 0 - 100 per section. High score = better quality of life.
EQ-5D-5L | 6 weeks, 6 months, 12 months
  Quality of life measure. Scored 0 - 100 for VAS. High score = better quality of life.
Walking distance | 6 weeks, 6 months, 12 months
  Walking distance, metres, self-reported.

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, PhD, Study Chair — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, UK, United Kingdom

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829